CLINICAL TRIAL: NCT05978778
Title: Effects of Active Video Gaming on Pre-handwriting Skills of Children With Down Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0722
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Effects of active video gaming on pre-handwriting skills of children with down's
  syndrome.
Who Masked: Participant
Masking Description: Effects of active video gaming on pre-handwriting skills of children with down's
  syndrome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (Other): Nine children will be randomly allocated to control group who receive only pre-hand writing skills.
  Interventions: Other: pre-hand writing skills
- Experimental group (Experimental): Nine children will be randomly allocated to experimental group who receive active video gaming along with pre-hand writing skills.
  Interventions: Device: wii sports game; Other: pre-hand writing skills

INTERVENTIONS:
Device: wii sports game — wii sports is a collection five sports game stimulation,which have been designed to demonstrate the motion sensing capabilities of wii remote
  Other Names: video gaming
  Arms: Experimental group
Other: pre-hand writing skills — pre-hand writing skills

SUMMARY:
Down's syndrome is a genetic disorder caused by trisomy 21. Down's syndrome is most common genetic mental disability that affects children physically, mentally and functionally. It occurs due to an extra copy of chromosome 21. It involves a slightly flattened facial profile, low muscle tone upward-slanted eyes, and ligamentous laxity. Central hypotonia, mental retardation and short stature are very common features of children with down's syndrome. Children with down's syndrome are characterized by awkward movements, gait, increased flexibility of joints, timing of mastering of basic skills and , under-development of fine motor skills. Active video gaming used different games that involve interactive session that can enhance cortical recognition, motor learning and functional profile of children with DS. The objective of this study is to determine the effects of active video gaming on pre-hand writing skills of children with down's syndrome. This will be a RCT(Randomized Controlled Trial).The sample size was 18 and the study design was a case-control trial. The inclusion criteria are children with down syndrome age 6 to 12 years both male and female patients are randomly selected and children with poor pre-hand writing skills. And the exclusion criteria for this study is children with any other neurological condition like (epilepsy, instability of atlantoaxial joints, cardiac anomalies,) vision, and hearing loss. Two groups were randomly assigned and equally divided patients into each group. Group A received pre-handwriting skills, like tracing alphabets and numbers, scribbling, coloring, painting, and group B received active video gaming and prehandwriting skills. For measuring each group developmental coordination

disorder questionnaire tool is used. The session will be taken 30 mins thrice a week for (8consecutive weeks). Data collected from different centers, Raising sun institute of special education. Autism resource center Lahore. SPSS for Windows software, version 25 will be used to analyze the data using statistical Significance p=0.05. The Shapiro-Wilk test will be used to check the normality of data. Keywords: Active video gaming, Down syndrome, Computer game, Fine motor skills, Pre-hand writing skills, Virtual reality gaming.

DETAILED DESCRIPTION:
To determine the effects of active video gaming on pre-hand writing skills of children with down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 to 14 years.
* Both male and female patient diagnosed with down syndrome.
* Able to understand and follow verbal command.
* Down syndrome children with pre-hand writing skills are not good.
* Difficulty in fine motor skills.

Exclusion Criteria:

* Patients will have any neurological sign (epilepsy, instability of the atlantoaxial joint, cardiac anomalies, vision and hearing loss, speech loss.
* Musculoskeletal and mobility disorder.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
pre handwriting skills syndrome. | 6 months
  bilateral hand use will determine by box and ball test children with down syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Nageen Zahra, ms, Principal Investigator — Ripha International Univerity
Locations (1):
- Lingua Speech Model town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'BRIEN JC, O'BRIEN MO. Educational Systems. Pediatric Skills for Occupational Therapy Assistants E-Book. 2020 Jul 12:46.